CLINICAL TRIAL: NCT02326870
Title: Evaluation of the Follow me Mode of the AutoLap System - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.S.T. Medical Surgery Technology LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AL-65-003
Record Dates: First submitted 2014-12-21; First posted 2014-12-30 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Patients Who Were Scheduled for General and Gynecological Laparoscopic Procedures
Keywords: laparoscopic Cholecystectomy; laparoscope holder; gynecological laparoscopy procedures; fundoplication surgery; laparoscopic adnexal surgery; excision of endometriosis lesion; diagnostic laparoscopy procedures; right hemicolectomy; Diaphragmatic hernia
MeSH Terms: conditions — Hernia, Diaphragmatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The AutoLap system (Experimental): Use of the AutoLap system for controlling the laparoscope during the procedure
  Interventions: Device: AutoLap

INTERVENTIONS:
Device: AutoLap

SUMMARY:
The main objectives of this study are to evaluate the performance and ease of use of the Follow me mode of the AutoLap system during general and gynecological laparoscopic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (ICF).
2. Patients over 18 years

Exclusion Criteria:

1. Pregnancy
2. Extensive adhesions that will preclude routine laparoscopic surgical approach.
3. American Society of Anesthesiologists' (ASA) classification>2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of successful "Follow Me" movements | during surgery
System set-up time | during surgery
Length of procedure | during surgery
Number of times that the laparoscope was removed for cleaning | during surgery
AutoLap evaluation questionnaire | post surgery

SECONDARY OUTCOMES:
System repositioning | during surgery

OTHER OUTCOMES:
Surgeon's learning curve for the use of the AutoLap system | post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Ivo A. M. J. Broeders, MD, Principal Investigator — Meander Medisch Centrum
Locations (4):
- Israel (2):
  - Assuta Medical Center, Haifa
  - Assuta Medical Center, Tel Aviv
- Netherlands (2):
  - Meander Medisch Centrum, Amersfoort
  - University Medical Center Utrecht, Utrecht